CLINICAL TRIAL: NCT01280331
Title: A Randomized, Double-Blind, Multi-Center, Repeat-Dose, Comparison of the Effects of Q8003 to the Morphine-Equivalent Doses of Oxycodone and of Morphine on the Opioid-Related Adverse Events of Moderate to Severe Nausea, Emesis, and Dizziness in Subjects With Acute Moderate-to-Severe Postoperative Pain Following Bunionectomy Surgery
Brief Title: Comparison of the Safety of Q8003 Versus Morphine Equivalent Doses of Its Components (Oxycodone and Morphine) in Bunionectomy Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: QRxPharma Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Q8003-022
Record Dates: First submitted 2011-01-18; First posted 2011-01-20 (Estimated); Last update posted 2012-05-17 (Estimated); Status verified 2012-05

CONDITIONS: Postoperative Pain
Keywords: Bunionectomy
MeSH Terms: conditions — Pain, Postoperative | interventions — MoxDuo; Morphine; Oxycodone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Q8003 12 mg/8 mg (Experimental): Combination
  Interventions: Drug: Q8003 (morphine sulfate and oxycodone hydrochloride)
- Morphine sulfate 24 mg (Active Comparator): Single component
  Interventions: Drug: Morphine sulfate
- Oxycodone HCl 16 mg (Active Comparator): Single component
  Interventions: Drug: Oxycodone HCl

INTERVENTIONS:
Drug: Q8003 (morphine sulfate and oxycodone hydrochloride) — Two Q8003 6 mg/4 mg IR Capsules q6h
  Arms: Q8003 12 mg/8 mg
Drug: Morphine sulfate — Two morphine sulfate 12 mg IR capsules q6h
  Arms: Morphine sulfate 24 mg
Drug: Oxycodone HCl — Two oxycodone HCl 8 mg IR Capsules q6h
  Arms: Oxycodone HCl 16 mg

SUMMARY:
This is a randomized, double-blind, multicenter, repeat-dose study of fixed doses of Q8003 12 mg/8 mg given q6hr compared to morphine sulfate 24 mg and oxycodone hydrochloride 16 mg given q6hr for the management of acute moderate to severe postoperative pain for 48 hours following bunionectomy surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patient is male or female and at least 18 years of age.
* Females must be non-pregnant, non-lactating, and practicing an acceptable method of birth control, or be surgically sterile or postmenopausal (amenorrhea for ≥ 12 months). Non-pregnancy will be confirmed by pregnancy tests conducted at Screening and Pre-treatment.
* Patient is scheduled for bunionectomy surgery, meets the criteria of an ASA Class I to III, and is willing to stay in the study center for at least 48 hours from the initial dose of study medication post surgery.
* To be randomized after surgery, the patient must report moderate to severe pain (a score of 2 or more on the 4 point Likert scale or 4 or more on the 11 point NPRS scale).
* At least 40% of study subjects will be 60 years of age or older.

Exclusion Criteria:

* In the opinion of the Investigator, has a history of pulmonary, cardiovascular (including uncontrolled hypertension), neurologic, endocrine, hepatic, gastrointestinal, or kidney disease or therapy that would jeopardize the patient's well being by participation in this study or is mentally or emotionally unsuitable to participate, or unable/unwilling to comply with the study assessments.
* Used opiates continuously (including tramadol) for more than ten days in the past year.
* Hypersensitivity or poor tolerance to acetaminophen.
* Currently receiving any medications that are not at a stable dose (the same dose for > 2 months prior to date of surgery).
* Was dosed with another investigational drug within 30 days prior to the Screening Visit or has previously received treatment with Q8003.
* Current therapy with central nervous system depressant medications that might increase the risks of treatment with opioids (other than those used with surgical anesthesia).
* Current evidence of alcohol abuse (regularly drinks more than 4 units of alcohol per day; 1 unit = ½ pint of beer, 1 glass of wine, or 1 ounce of spirit).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 375 (Actual)
Dates: Start 2011-01; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
Differences in desaturation events per standardized time unit | 48 hours

SECONDARY OUTCOMES:
Difference in efficacy between Q8003 and its components (morphine and oxycodone) | 48 hours
  Changes from baseline in pain intensity
Differences in the absence of emesis without the use of an anti-emetic (emesis complete response) | 48 hours

CONTACTS AND LOCATIONS:
Overall Officials: Patricia T. Richards, MD, Ph.D., Study Director — QRxPharma Inc.
Locations (4):
- United States (4):
  - Investigational site, Anaheim, California
  - Investigational site, Owings Mills, Maryland
  - Investigational site, Pasadena, Maryland
  - Investigational Site, San Antonio, Texas